CLINICAL TRIAL: NCT06241612
Title: Individualized Elective Neck Irradiation Based on the Lymph Node Metastasis Pattern in NPC Patients
Brief Title: Individualized Elective Neck Irradiation in NPC Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First People's Hospital of Foshan (Other); Sichuan Cancer Hospital and Research Institute (Other); Xiangya Hospital of Central South University (Other); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); Eye & ENT Hospital of Fudan University (Other); First Affiliated Hospital of Guangxi Medical University (Other); First Hospital of China Medical University (Other); Renmin Hospital of Wuhan University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Qingyuan People's Hospital (Other)
Responsible Party: Principal Investigator, Ling-Long Tang, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2023-651-01
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard group (Active Comparator): Upper-neck irradiation at the uninvolved neck
  Interventions: Radiation: Individualized Elective Neck Irradiation
- Experimental group (Experimental): The low-risk clinical target volume would be reduced to two vertebral levels below the vertebral level of the metastatic level II-V nodes.
  Interventions: Radiation: Individualized Elective Neck Irradiation

INTERVENTIONS:
Radiation: Individualized Elective Neck Irradiation — Individualized Elective Neck Irradiation

SUMMARY:
To evaluate whether individualized elective neck irradiation for nasopharyngeal carcinoma based on the vertebral level of metastatic lymph nodes can reduce the incidence of radiation-related adverse effects and improve patients' quality of life，without reducing survival.

DETAILED DESCRIPTION:
A multicenter phase III noninferiority randomized trial (NCT02642107) showed that upper-neck irradiation at the uninvolved neck resulted in comparable regional control and survival rate to standard whole-neck irradiation in NPC, reduced late toxicity of hypothyroidism, dysphagia, and neck tissue damage, and improved quality of life, including fatigue and swallowing.

However, the vertical range of the upper neck is extensive, necessitating further reduction in the scope of prophylactic irradiation. By integrating MRI and PET-CT to accurately assess metastatic lymph nodes and their corresponding vertebral levels, the investigators identified a pattern of sequential lymph node metastasis descending along the vertebral body in the vertical direction. Further correlative analysis revealed that nodal metastasis at any one of the vertebral levels strongly and positively correlated with metastasis at two adjacent vertebral levels, including one level above and one below.

Considering this, the investigators propose the following scientific hypothesis: individualized elective neck irradiation for nasopharyngeal carcinoma based on the vertebral level of metastatic lymph nodes can reduce the incidence of radiation-related adverse effects and improve patients' quality of life, without reducing survival. The investigators thus conduct a multicenter randomized phase 3 trial to verify their hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* The eligibility criteria are: newly diagnosed, untreated, non-distant metastatic, and non-keratinizing NPC; nodes are diagnosed with PET/CT and MRI; staged as T1-4N0-2 or N3 category of non-bilateral lower-neck node metastasis; aged between 18 and 70 years; Karnofsky performance-status score > 70; adequate haematological function, with a leucocyte count > 4 × 109/L, haemoglobin > 90 g/L, and a thrombocyte count > 100×109/L

Exclusion Criteria:

* The exclusion criteria include: previous chemotherapy treatment, surgery (except diagnostic) or radiotherapy to the neck or nasopharyngeal regions; previous malignancy; lactation or pregnancy; or severe coexisting illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Regional relapse-free survival | 3 years
  The regional relapse-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to the date of nodal relapse or death from any cause, whichever occurred first. Their differences will be compared between treatment arms using the log-rank test.

SECONDARY OUTCOMES:
Radiation-related toxicity | Within 3 month after radiotherapy for acute toxicity; long term for late toxicity
  Acute and late toxicity will be documented according to RTOG/EORTC System and the CTCAE(Common Terminology Criteria for Adverse Events). Toxicity will be summarized using descriptive statistics.
Overall survival | 3 years
  The overall survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to death from any cause. Their differences will be compared between treatment arms using the log-rank test.
Local relapse-free survival | 3 years
  The local relapse-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to documented local relapse or death from any cause. Their differences will be compared between treatment arms using the log-rank test.
Distant metastasis-free survival | 3 years
  The distant metastasis-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to documented distant metastasis or death from any cause. Their differences will be compared between treatment arms using the log-rank test.
Patient's quality-of-life: global health status | 3 years
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on global health status suggest better health.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No